CLINICAL TRIAL: NCT00397098
Title: A Double-Blind Randomized Withdrawal Study Evaluating the Efficacy and Safety of SR58611A Versus Placebo in the Prevention of Relapse of Anxiety up to 1 Year in Patients With GAD Improved After 12 Weeks of Open Label Treatment With SR58611A.
Brief Title: Prevention of Relapse Study of SR58611A in Improved Patients With Generalized Anxiety Disorder
Acronym: VEGA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: reprioritization of indications
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTE5894; EudraCT 2006-002253-71
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Anxiety Disorders
Keywords: Anxiety disorders, Relapse prevention
MeSH Terms: conditions — Anxiety Disorders | interventions — Amibegron hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SR58611A

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of SR58611A (350 mg BID) compared to placebo in the prevention of relapse of anxiety, in patients with Generalized Anxiety Disorder improved after 12 weeks of treatment with SR58611A.

The primary objective is to evaluate the efficacy of SR58611A 350mg BID compared to placebo over a 24 to 52-week treatment period.

The secondary objective is to assess the safety and tolerability of SR58611A in patients with GAD.

ELIGIBILITY:
Inclusion Criteria:

For entry into the open phase:

* Patients suffering from generalized anxiety disorder, according to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) criteria and assessed with the Mini International Neuropsychiatric Interview (MINI) plus Generalized Anxiety Disorder (GAD) module.
* With a total score on the 14-item Hamilton Anxiety Rating Scale (HAM-A) > 20 at V1(D-4) and V2 (D-1).

For entry into the double-blind randomized phase:

* Improved patients with HAM-A score < 11 at V7 (W12).

Exclusion Criteria:

* Inpatients.
* Patients with a diagnosis of Major Depressive Disorder (DSM IV-TR) within 6 months of screening.
* Patients with a MADRS total score > 18 at screening or baseline.
* Patients at immediate risk for suicidal behaviour.
* Patients with other current (within 6 months) anxiety disorder according to the MINI
* Patients with a lifetime history according to the MINI of: Bipolar disorder, Psychotic disorder, Antisocial personality disorder.
* Patients with a current history according to the MINI of: Anorexia nervosa or bulimia nervosa in the past 6 months, Alcohol or substance dependence or abuse in the past 12 months, except nicotine or caffeine dependence.

The investigator will evaluate whether there are other reasons why a patient may not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2006-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary criterion is the time to relapse of anxious symptoms (in days) from randomization date defined by either:
HAM-A total score ≥ 15 confirmed at a subsequent visit 2 weeks later unless the patient drops out,or
Any drop-out for lack of efficacy (according to investigator's decision),or
Prescription/use of alternative or additional treatments for relief of psychiatric symptoms.

SECONDARY OUTCOMES:
Change from baseline (V7) in:-Clinical Global Impression (CGI) Severity of Illness Score
Hamilton Anxiety Rating Scale (HAM-A)

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (9):
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Barcelona, Spain

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com